CLINICAL TRIAL: NCT02921750
Title: A Randomised Multi-centre Non-inferiority Investigation to Evaluate the Efficacy and Safety of Exufiber Versus Aquacel Extra in Moderately or Strongly Exuding Venous and Mixed Ulcers of Predominantly Venous Origin
Brief Title: Investigation to Evaluate the Efficacy and Safety of Exufiber Versus Aquacel Extra in Moderately or Strongly Exuding Venous and Mixed Ulcers of Predominantly Venous Origin
Acronym: PD-497314
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEXU03
Record Dates: First submitted 2016-09-19; First posted 2016-10-03 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Venous Leg Ulcer
Keywords: wound reduction wound healing, venous ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dressing Exufiber®Gelling Fibre Dressing (Experimental): will receive dressing Exufiber®
  Interventions: Device: Exufiber Gelling Fibre Dressing
- Dressing Aquacel®ExtraHydrofiber®Dressing with Strengthenin (Active Comparator): Will receive Aquacel®Extra™
  Interventions: Device: Aquacel Extra Hydrofiber® Dressing with Strengthening Fibre

INTERVENTIONS:
Device: Exufiber Gelling Fibre Dressing — Gelling fibre dressing
  Arms: Dressing Exufiber®Gelling Fibre Dressing
Device: Aquacel Extra Hydrofiber® Dressing with Strengthening Fibre — Hydrofiber® Dressing with Strengthening Fibre
  Arms: Dressing Aquacel®ExtraHydrofiber®Dressing with Strengthenin

SUMMARY:
The investigation is designed as an open, randomized, non-inferiority, multi-centre investigation.

212 evaluable subjects will be randomised. Subjects to be included will suffer from an exuding venous or mixed ulcer of predominantly venous origin. Subjects will either be randomized to Exufiber®Gelling Fibre Dressing or Aquacel®Extra Hydrofiber® Dressing with Strengthening Fibre using, centralized randomization

DETAILED DESCRIPTION:
Visits are planned for baseline followed by 1, 2, 3, 4 and 6 weeks post treatment. The sub-group of at least 50 subjects will also be followed at week 8, 12, 16, 20, and 24 post treatment or until wound is healed if earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent i.e. subject must be able to understand and sign the Patient Information and Consent Form
2. Both gender ≥18 years old
3. Ulcer moderately or strongly exudative justifying the use of an absorbent dressing
4. (History of compression at least two weeks before inclusion) Deleted in Am.2
5. (Wound covered with slough ≥70%) Deleted in Am.4
6. 0.7≤ABPI<1.3
7. Ulcer duration 6 weeks to 60 months
8. Ulcer size 3 cm2-100 cm2
9. Target ulcer at least 3 cm away from any other lesion

Exclusion Criteria:

1. Known allergy/hypersensitivity to the dressings
2. Pregnant or breastfeeding
3. Circumferential wounds (the entire wound should be able to be captured on a single image/photo)
4. Subjects who will have problems following the protocol
5. Subjects included in other ongoing clinical investigation evaluating wound dressings at present or during the past 30 days
6. Patient with a systemic infection not controlled by suitable antibiotic treatment
7. Clinically infected wound according to the judgement of the investigator (heat, pain, swelling, redness or purulent secretion)
8. Wound covered with black necrosis
9. Dry wounds
10. Malignant wound degeneration
11. Current treatment with radiotherapy, chemotherapy, immunosuppressant drugs or high doses of oral corticosteroids if any
12. Subject with deep vein thrombosis within 3 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Joergensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (33):
- Czechia (7):
  - St. Ann University Hospital Dep of Dermatovenereology, Brno
  - Hospital Jihlava, Jihlava
  - Regional hospital Pardubice Dermatology Department, Pardubice
  - Fakultní nemocnice Královské Vinohrady (FNKV)Department of General Surgery 3, Prague
  - General University Hospital in Prague, Prague
  - Diabetologie, Soběslav
  - Salvatella LTD, Třinec
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark
- France (6):
  - Hôpital Michallon, Grenoble
  - Groupe Hospitalier, La Rochelle
  - Hospital Géneral du Mans, Le Mans
  - Clinique du Parc Unité de Cicatrisation, Lyon
  - CHU Nantes, Nantes
  - Clinique Pasteur, Toulouse
- Germany (10):
  - Wundzentrum Augsburg, Augsburg
  - WundZentrum Dortmund, Dortmund
  - WundZentrum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Venenzentrum Freiburg, Freiburg im Breisgau
  - Paracelsus-Klinik am Silbersee, Hanover
  - University Hospital Schleswig-Holstein, Kiel
  - Johannes-Gutenberg-Universität Mainz, Mainz
  - WundZentrum München Nord, München
  - WundZentrum Ulm, Ulm
- Poland (4):
  - Usługi Medyczne PRO-MED Sp. z o.o., ul., Gliwice
  - Niepubliczny Zakład Opieki Zdrowotnej "GAM-MED", ul., Kielce
  - Niepubliczny Zakład Opieki Zdrowotnej "Mikomed", ul., Lodz
  - Medical Hair & Esthetic, ul., Lublin
- Sweden (5):
  - Lund university Hospital,, Lund
  - Avdelningen för kliniska prövningar, Universitetssjukhuset Örebro, Örebro
  - Skellefteå Lasarett, Skellefteå
  - Karolinska Trial Alliance, Prim, Stockholm
  - Södersjukhuset (Sårcentrum), Stockholm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exufiber: Investigational Device: Exufiber® gelling fibre dressing as primary dressing to facilitate moist healing of venous leg ulcer.
- Aquacel: Comparator - Aquacel® Extra™ Hydrofiber® Dressing with Strengthening Fibre as primary dressing to facilitate moist healing of venous leg ulcer.
Period: Overall Study
Arm/Group | Exufiber | Aquacel
Started (Safety population) | 124 | 124
Intention to Treat (ITT) | 122 | 123
Per Protocol (PP) | 100 | 107
Completed 6 Weeks Follow-up (PP) | 97 | 104
Subgroup Followed for 24 Weeks (ITT) | 35 | 40
Subgroup Followed for 24 Weeks (PP) | 19 | 36
Completed (Completed 6 weeks follow-up) | 115 | 113
Not Completed | 9 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Wound healed | 3 | 3
Not completed — Serious Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Exufiber: Investigational device: Exufiber Gelling fibre dressing
- Aquacel: Comparator: Aquacel® Extra™ Hydrofiber® Dressing with Strengthening Fibre
- Total: Total of all reporting groups
Arm/Group | Exufiber | Aquacel | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 47 | 88
  >=65 years | 81 | 76 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (12.3) | 69.0 (15.0) | 69.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 69 | 131
  Male | 60 | 54 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 89 | 93 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 30 | 63
Region of Enrollment [Number; unit: participants] — Population: Intention to treat population
  participants
    Czechia: number analyzed (Participants) | 17 | 21 | 38
    Czechia | 17 | 21 | 38
    Denmark: number analyzed (Participants) | 3 | 6 | 9
    Denmark | 3 | 6 | 9
    Poland: number analyzed (Participants) | 48 | 51 | 99
    Poland | 48 | 51 | 99
    France: number analyzed (Participants) | 21 | 25 | 46
    France | 21 | 25 | 46
    Germany: number analyzed (Participants) | 18 | 15 | 33
    Germany | 18 | 15 | 33
    Sweden: number analyzed (Participants) | 15 | 5 | 20
    Sweden | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Wound Area Change (%)
Description: The primary endpoint was to measure relative reduction of wound area (%) from baseline to end of investigation (up to 6 weeks measured by the validated system PictZar on the photos taken after debridement at week 0, week 4, and week 6 (or final visit if healed earlier)
Time Frame: 6 weeks
Population: PP analysis set, tested for non-inferiority
Measure: Median (Full Range); unit: relative wound area change in percentage
Groups:
- Exufiber: Investigational device, Exufiber Gelling Fibre Dressing
- Aquacel: Comparator, Aquacel® Extra™ Hydrofiber® dressing with strengthening fibre
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 100 | 107
relative wound area change in percentage | -49.7 [-100 to 191.2] | -42.4 [-100 to 1538.4]
Statistical Analysis 1: Comparison: Exufiber vs Aquacel; Test type: Non-Inferiority — In this non-inferiority study the primary efficacy analysis included constructing a two sided 95% confidence interval, using Fisher's non-parametric permutation test, for between-treatment differences (Exufiber - Aquacel Extra) in the mean percentage area change from baseline to 6 weeks. This means that if the lower limit of this confidence interval was found to be greater than 12%, non-inferiority will be established; p = 0.093, Fisher Exact; Mean Difference (Final Values) = -29.4, 95% CI 2-sided [-63.5 to 3.2]

2. Secondary Outcome: Wound Area Change (cm2)
Description: The secondary endpoint was to measure relative reduction of wound area (cm2) from baseline to end of investigation (up to 6 weeks measured by the validated system PictZar on the photos taken after debridement at week 0, week 4, and week 6 (or final visit if healed earlier)
Time Frame: 6 weeks
Population: ITT analysis set
Measure: Mean (Standard Deviation); unit: relative wound area change in cm2
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
relative wound area change in cm2 | -4.64 (7.73) | -3.48 (7.59)

3. Secondary Outcome: Linear Advance of Wound Margin
Description: Linear advance of the wound margin according to Gilman's formula (G= [(A0-An) / ((P0+Pn) / 2)] / Time) was calculated and evaluated using the validated system PictZar on the photos taken after debridement. The values represent wound margin advanced inwards over time (i.e., reduction in perimeter) presented in cm/day.
Time Frame: 6 weeks
Population: ITT analysis set.
Measure: Mean (Standard Deviation); unit: cm/day
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
cm/day | 0.008 (0.010) | 0.007 (0.010)

4. Secondary Outcome: Pain During Debridement
Description: Pain was reported by patients and measured by Visual Analogue Scale (VAS) 0-100mm, where 0=is no pain, 100=is worst pain ever.
Time Frame: 6 weeks
Population: ITT analysis set
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
mm | 25.8 (27.2) | 26.9 (29.0)

5. Secondary Outcome: Pain at Dressing Removal
Description: as for outcome 4
Time Frame: 6 weeks
Population: ITT analysis set
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
mm | 16.3 (22.0) | 16.9 (22.8)

6. Secondary Outcome: Percentage of Clinicians of Opinion 'Very Good' for Dressing Features
Description: Clinician reported outcomed by means a questionnaire was used to capture opinions related to the two dressing types. Reply alternatives varied between very poor, poor, good, very good. Results reported as 'very good' are presented as a percentage based on all follow-up visits aggregated.
Time Frame: 6 weeks
Population: ITT analysis set.
Measure: Number; unit: Percentage reported 'very good'
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
Percentage reported 'very good'
  Ease of application of dressing | 58.4 | 57.5
  Ease of removal of dressing | 48.7 | 35.9
  Flexibility of dressing | 48.0 | 40.8
  Overall experience of dressing | 46 | 32.5
  Conformability to the wound | 39.9 | 36.2
  Ability to Absorb Exudates | 49.2 | 32.3
  Ability to Retain Exudate | 47.8 | 31.7
  Ability to Absorb Blood | 38.4 | 32.5
  Ability to Keep Blood and Slough | 36.3 | 28.1

7. Secondary Outcome: Percentage of Clinicians of Opinion 'Does Not Adhere' Related to Dressing Features
Description: Clinician reported outcomed by means a questionnaire was used to capture opinions related to the two dressing types. Reply alternatives varied between does not adhere, adhere a little, adhere a lot. Results reported as 'does not adhere' are presented as a percentage based on all follow-up visits aggregated.
Time Frame: 6 weeks
Population: ITT analysis set.
Measure: Number; unit: Percentage reported 'does not adhere'
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 122 | 123
Percentage reported 'does not adhere'
  Non-adherence to wound bed at removal | 44.2 | 31.1
  Non-adherence to peri-wound skin at removal | 72.0 | 52.1

8. Other Pre Specified Outcome: Percentage of Participants With Healed Wounds
Description: Wound healing assessments were based on blind independent clinical review of photos.
Time Frame: from baseline to 24 weeks
Population: Subgroup followed until healing or up to 24 weeks.
Measure: Number; unit: Percentage of participants
Groups:
- Aquacel: Comparator Aquacel® Extra™ Hydrofiber® dressing with strengthening fibre
Arm/Group | Exufiber | Aquacel
Number analyzed (Participants) | 35 | 40
Percentage of participants | 40.0 | 47.5

ADVERSE EVENTS:
Time Frame: Adverse event were collected while subjects participated in the study, i.e. from the baseline visit, to 6 or 24 weeks follow-up, or until wound healing/premature study termination. h
Arm/Group | Exufiber | Aquacel
All-Cause Mortality (participants affected / at risk) | 1/124 | 1/124
Serious Adverse Events (participants affected / at risk) | 5/124 | 8/124
Other Adverse Events (participants affected / at risk) | 18/124 | 19/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exufiber (N=124) | Aquacel (N=124)
Fracture and hospitalisation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient was fallen down and broke her left arm. Of Cause of that she needs an Operation and was in hospital.
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Erysipelas right leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastric hemorrhage with hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (Renal and urinary disorders) | 1 (1) | 1 (1) — Death unknown cause in the Aquacel group. Death due to acute renal failure in the Exufiber group
Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient has increase pain, the wound status is going worse
Infection exacerbated COPD (Renal and urinary disorders) | 0 (0) | 1 (1)
Erysipelas PDK, hospitalize (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intensification of depression (Psychiatric disorders) | 0 (0) | 1 (1) — Intensification of depression symptoms in course of schizophrenia
Circulatory insufficiency with dehydration and dizziness (General disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exufiber (N=124) | Aquacel (N=124)
Skin reaction around the wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Severe irritation around the wound. The dressing was done every 2 days with 2 Aquacel on the wound, contrary to the instructions of the protocol (a daily frequency with only 1 AQUACEL on the wound).
Scheduled hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Infection at study wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound infection right leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Wound infection right leg, and Increased redness in peri-wound skin.
Increased wound liquid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The wound was covered with lots of blue-green-coloured slough, which Looks like pseudomonas
Skin blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Small skin blister and wound on the leg at the at area of dressing tape
Aggravation of known psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Strong itching in the marginal area of the wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection of the target ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall at home with wound in the right leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache, tiredness (General disorders) | 0 (0) | 1 (1)
Cough and inceased temperature (Infections and infestations) | 0 (0) | 1 (1)
Erysipel of nonstudy leg - left leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Burning, erhema of the scalp. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Aquacel dressing intolerance (burn and redness) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increasing the ulcer with inflammatory reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
New ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Local infection in study wound (Infections and infestations) | 2 (2) | 0 (0)
Periwound skin irritation and blistering in study wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flu infectious for 3 weeks (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Redness and irritation on Periwound Skin on left leg study ulcer . (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swollen right ankle/foot. (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ulcer exacerbation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stinging or burning while wearing study product (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Local signs of infection at the target wound (Infections and infestations) | 1 (1) | 0 (0)
Eczema with tingling and pain on right foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain in back due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Pain of the wound unrelated to the dressing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02921750/SAP_000.pdf
  • Study Protocol (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT02921750/Prot_001.pdf